CLINICAL TRIAL: NCT01359137
Title: An Assessment of Arizona's SAFE (Swift Accountable Fair Enforcement) Program in Cochise County
Brief Title: An Assessment of SAFE (Swift Accountable Fair Enforcement) in Cochise County
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pepperdine University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPP0311F09
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Behavior
Keywords: Behavior; Drug users; Criminal Justice; Probation
MeSH Terms: conditions — Behavior; Drug Misuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probation as usual (Experimental): Routine supervision with no deferred jail condition.
  Interventions: Behavioral: Probation as usual
- Deferred jail (Experimental): Discretionary deferred jail in response to violations of probation conditions.
  Interventions: Behavioral: Deferred Jail
- Arizona's SAFE (Experimental): Swift Accountable Fair Enforcement (SAFE) which uses non-discretionary brief jail sanctions for probation violations.
  Interventions: Behavioral: Arizona's SAFE

INTERVENTIONS:
Behavioral: Probation as usual — Routine probation with do deferred jail condition.
  Other Names: PAU
  Arms: Probation as usual
Behavioral: Deferred Jail — Discretionary deferred jail in response to violations of probation conditions.
  Other Names: DIS
  Arms: Deferred jail
Behavioral: Arizona's SAFE — Swift Accountable Fair Enforcement (SAFE) uses non-discretionary brief jail sanctions for probation violations.
  Other Names: Swift Accountable Fair Enforcement; HOPE
  Arms: Arizona's SAFE

SUMMARY:
This is a Cochise County experiment with innovative probation supervision practices. Subjects are assigned to one of three supervision conditions.

DETAILED DESCRIPTION:
Historically, rates of failure on routine probation have been high. The result is that large numbers of probationers are ultimately revoked from probation and sentenced to long underlying jail or prison terms. Arizona is experimenting with alternatives to routine probation with the goal of reducing the overall burden of incarceration. Cochise County in Arizona is experimenting with innovative probation supervision practices. Subjects are assigned to one of three supervision conditions: Probation-as-usual (routine supervision with no deferred jail); discretionary deferred jail in response to probation violations; and Arizona's Swift, Accountable, Fair, Enforcement, or SAFE (SAFE involves non-discretionary deferred jail in response to probation violations).

ELIGIBILITY:
Inclusion Criteria:

* Supervised on probation in Cochise County
* Residing in Cochise County

Exclusion Criteria:

* First-time marijuana possession cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Revocation rate | 12 months
  Percentage of subjects in each condition who are revoked from probation and returned to jail or prison.

SECONDARY OUTCOMES:
% positive drug tests | 12 months
  Percentage of random and scheduled drug tests that test positive for illicit drugs
Days incarcerated | 12 months
  Total number of days incarcerated in jail and prison
% Missed appointments | 12 months
  Percentage of probation appointments that are missed
New arrests | 12 months
  Number of new arrests

CONTACTS AND LOCATIONS:
Locations (1):
- Cochise County Adult Probation Department, Bisbee, Arizona, United States